CLINICAL TRIAL: NCT03781232
Title: Non-invasive Glucose Measurement With Raman Technology. Calibration of Newly Developed Devices in Patients With Type 1 and Type 2 Diabetes - Glucobrunn Study
Brief Title: Non-invasive Glucose Measurement With Raman Technology in Patients With Type 1 and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RSP-09
Record Dates: First submitted 2018-11-21; First posted 2018-12-19 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Diabete Mellitus; Medical Device
Keywords: Non-invasive glucose monitoring; Raman spectroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSP-09-01 (Experimental): Enrolled subjects will perform 4 daily measurement session during their regular stay at the clinic. A measurement session consists of a reference capillary blood sample and two measurements on the Prototype 0.3.
  Interventions: Device: Prototype 0.3
- RSP-09-02 (Experimental): Enrolled subjects will measure at home for 26 six days and visit the clinic two times. During home measurements, 6 measurement sessions will be performed by the subject a day. A measurement session consists of two BGMs, two CGMs and two measurements on the Prototype 0.3. On in-clinic visits the subject will be administered a high glucose breakfast and the following 6-7 hours, measurement sessions will be performed every 15 minutes.
  Interventions: Device: Prototype 0.3

INTERVENTIONS:
Device: Prototype 0.3 — Prototype 0.3 is a non-invasive glucose monitoring device using Raman spectroscopy

SUMMARY:
The study was established to collect data and reference measurements in order to establish calibration models for the Prototype 0.3

DETAILED DESCRIPTION:
Subjects are recruited at two different sites.

Site 1: In group 1 subjects will on their regular stay in the clinic perform four measurement sessions a day. A measurement session consist of a reference capillary blood sample and two measures on the IMD.

Site 2: The study in group 2 consists of 26 home-based measurements and two in-clinic days. During the home measurements, 6 measurement sessions will be performed by the subjects a day. A measurement session consists of two reference BGMs, two reference CGMs and two measurements on the device. On in-clinic visits, subjects will be administered high glucose breakfast and the following 6-7 hours, measurement sessions are performed every 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Have a diagnosis of type 1 or type 2 diabetes mellitus (for RSP-09-02, only patients with type 1 diabetes)
* Skin phototype 1-4
* Be willing to perform a minimum of 6 / 12 (31 during excursion days) finger sticks per day during the study
* Be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol
* Be willing to provide written signed and dated informed consent

Exclusion Criteria:

* Inability to comply with the study procedures as described by the study protocol, according to the opinion of the investigator, due to e.g. known psychiatric diagnoses, lack of cognitive ability, alcohol dependency, drug use, psychosocial overload
* Have known severe allergy to medical grade adhesive or isopropyl alcohol used to clean the skin
* Be breastfeeding, pregnant, attempting to conceive or not willing and able to practice birth control during the study execution (applicable to female subjects only)
* Unable to hold hand/arm steadily (including tremors and Parkinson's Disease)
* Severe diabetes related complications such as advanced autonomic neuropathy, kidney disease, foot ulcers, legal blindness, or symptomatic cardiovascular disease as evidenced by a history of cardiovascular episode(s)
* Systemic or topical administration of glucocorticoids for the past 7 days
* Undergoing dialysis treatment
* Have extensive skin changes/diseases at the proposed measurement site (thenar) that could interfere with the accuracy of interstitial glucose measurements
* Have a concomitant medical condition which could interfere with the study devices (study arm 1: intake of acetaminophen study arm 2: intake of salicylic acid or higher doses of ascorbic acid)
* Unsuitable for participation due to any other cause as determined by the Investigator. Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation e.g. with required documentation
* Dependency from the sponsor or the clinical investigator (e.g. co-workers of the sponsor, the study site, and/ or their families)

Additional exclusion criteria for study arm 2:

* Severe hypoglycemia resulting in seizure or loss of consciousness in the 3 months prior to enrollment
* Hypoglycemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Generation and validation of predictive models by Inter Subject Unified Performance (ISUP). | 2 years
  Spectral Raman data will be collected together with paired reference measurements. Collected data will be used to generate calibration models capable of predicting tissue glucose levels.
  Models will be validated on independent data sets using the ISUP measure.
Generation and validation of predictive models by Mean Absolute Relative Difference (MARD) measures | 2 years
  Spectral Raman data will be collected together with paired reference measurements. Collected data will be used to generate calibration models capable of predicting tissue glucose levels.
  Models will be validated on independent data sets using the MARD measure.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Freckmann, Dr., Principal Investigator — Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm
Locations (2):
- Germany (2):
  - m&i-Fachklinik Bad Heilbrunn - Zentrum für Diabetes und Stoffwechselerkrankungen, Bad Heilbrunn
  - Institut für Diabetes-Technologie, Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No